CLINICAL TRIAL: NCT05618847
Title: Effects of Active Cycle of Breathing Technique With and Without Acapella on Airway Clearance, Dyspnea and Pulmonary Function Test in Chronic Obstructive Pulmonary Disease Patients
Brief Title: Effects of Active Cycle of Breathing Technique With and Without Acapella on Airway Clearance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC&Mishal Sabir
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: ACBT, Acapella, COPD, PEP
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active cycle of breathing technique with acapella (Experimental): Sit up with good posture to use the Acapella. Take in a fairly deep breath and hold it for about 3 seconds. Place the Acapella mouthpiece in your mouth. Seal your lips tightly around the mouthpiece.
  Exhale as much as possible (but not to forcefully) through the mouthpiece. Keep your cheeks as firm as possible when you exhale. Try not to inhale through the device.
  Repeat this maneuver for 10 breaths. Try to resist coughing during this phase. After these 10 blows, perform 3 huffs, then a big cough to bring the sputum up and out. Try not to swallow the mucus
  Interventions: Device: Acapella,ACBTS; Other: ACBTs
- active cycle of breathing technique (Active Comparator): Ask patient to breathe in and out gently through nose if he/she can. If patient breathe out through their mouth. Ask patient to let go of any tension in body with each breath out. Gradually try to make the breaths slower. Ask patient to take a long, slow, deep breath in, through nose. Try to keep chest and shoulders relaxed. Repeat 3-5 times. Huff is exhaling through an open mouth and throat instead of coughing. It helps move sputum up in airways so that patient can clear it in a controlled way. To 'huff' ask patient to squeeze air quickly from lungs, out through open mouth and throat, as if trying to mist up a mirror or glasses. Ask to use abdominal muscles to help squeeze the air out, but do not force it so much that cause wheezing or tightness in chest. Huffing should always be followed by breathing control.
  Interventions: Other: ACBTs

INTERVENTIONS:
Device: Acapella,ACBTS — Every subject will perform supervised ACBTs with and without acapella for four weeks. Three sessions per week will be given with 20 repetitions in two sets
  Arms: active cycle of breathing technique with acapella
Other: ACBTs — Every subject will perform supervised ACBTs with and without acapella for four weeks. Three sessions per week will be given with 20 repetitions in two sets

SUMMARY:
We are conducting this study to check the effects of active cycle of breathing technique with or without acapella on airway clearance, dyspnea and pulmonary function test in COPD patients.

Study design will be randomized controlled trial. Research will be conducted at Aziz Bhatti Shaheed Teaching Hospital and National Hospital Gujrat. Written informed consent will be obtained. Patients will be allocated randomly in two groups. Subjects will meet the predetermined inclusion and exclusion criteria. Questionnaire used as subjective measurements of dyspnea and sputum will be given and pulmonary function test values will be obtained prior to any intervention. One group will receive active cycle of breathing technique and the other group will receive active cycle of breathing technique with acapella device. Every subject will perform supervised ACBTs with and without acapella for four weeks. Three sessions per week will be given with 20 repetitions in two sets. At the end of 4 weeks treatment session, pulmonary function test values will be monitored and questionnaire will be obtained for dyspnea and sputum. Data will be analyzed on SPSS 25

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a non-communicable progressive and non-curable disease, characterized by persistent respiratory symptoms and airflow limitation. It is potentially fatal and it is the fourth cause of death in the world. Active Cycle of Breathing Techniques can be used to mobilize and clear excess pulmonary secretions and to generally improve lung function Loosen and clear secretions from the lungs. Three main phases of Active Cycle of Breathing Techniques are Breathing Control, Deep Breathing Exercises or Thoracic Expansion Exercises and Huffing or Forced Expiratory Technique. Acapella is a small hand held device for airway clearance. It has both resistive and vibratory features, which help to loosen and clear secretions from chest. This causes the vibration and resistance to the airflow which is then transmitted to the lungs. The resistance to the airflow will help to keep the airways open to get air behind the sputum and help it move upwards. The vibrations will help to loosen secretions from airways and move them up more easily for effective chest clearance. We are conducting this study to check the effects of active cycle of breathing technique with or without acapella on airway clearance, dyspnea and pulmonary function test in COPD patients.

Study design will be randomized controlled trial. Research will be conducted at Aziz Bhatti Shaheed Teaching Hospital and National Hospital Gujrat. Written informed consent will be obtained. Patients will be allocated randomly in two groups. Subjects will meet the predetermined inclusion and exclusion criteria. Questionnaire used as subjective measurements of dyspnea and sputum will be given and pulmonary function test values will be obtained prior to any intervention. One group will receive active cycle of breathing technique and the other group will receive active cycle of breathing technique with acapella device. Every subject will perform supervised ACBTs with and without acapella for four weeks. Three sessions per week will be given with 20 repetitions in two sets. At the end of 4 weeks treatment session, pulmonary function test values will be monitored and questionnaire will be obtained for dyspnea and sputum. Data will be analyzed on SPSS 25

ELIGIBILITY:
Inclusion Criteria:

* • Age:45-75

  * Both genders
  * Mentally stable
  * Diagnosed patients of COPD

Exclusion Criteria:

* • Any neurological condition

  * Arrythmias
  * Heart failure
  * Previous heart or lung surgery

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Sputum diary | 4 weeks
  The diary card has a graded symptom score for dyspnea, sputum volume and sputum color. In addition, the card includes a score for patient well-being and documented all minor symptoms (cough, chest pain, cold, or flu-like symptoms)
Dyspnea-MDP scale | 4 weeks
  The Multidimensional Dyspnea Profile (MDP) assesses overall breathing discomfort, sensory qualities, and emotional responses
Pulmonary function test | 4 weeks
  Pulmonary function tests (PFTS) are an important tool in the investigation and monitoring of patients with respiratory pathology. They provide important information relating to the large and small airways, the pulmonary parenchyma and the size and integrity of the pulmonary capillary bed

CONTACTS AND LOCATIONS:
Overall Officials: Madiha younas, MS, Principal Investigator — riphah internationl university
Locations (1):
- Aziz bhatti shaheed teaching hospital, Dhok Gujra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No